CLINICAL TRIAL: NCT00118716
Title: A Stratified, Multicenter, Randomized, Double-Blind, Parallel Group, 4-Week Comparison of Fluticasone Propionate/Salmeterol DISKUS Combination Product 100/50mcg BID Versus Fluticasone Propionate DISKUS 100mcg BID in Pediatric and Adolescent Subjects With Activity-Induced Bronchospasm
Brief Title: A Study Measuring Asthma Control In Pediatric And Adolescent Subjects Whose Asthma Is Worsened By Activity Or Exercise
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Purpose: Treatment
Other Study IDs: SFA100314
Record Dates: First submitted 2005-07-01; First posted 2005-07-12 (Estimated); Results first posted 2019-02-05 (Actual); Last update posted 2019-02-05 (Actual); Status verified 2017-12

CONDITIONS: Bronchospasm; Activity/Exercise Induced Bronchospasm
Keywords: asthma; bronchospasm
MeSH Terms: conditions — Bronchial Spasm; Motor Activity; Asthma, Exercise-Induced; Asthma | interventions — Fluticasone-Salmeterol Drug Combination; Fluticasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- FSC 100/50 mcg BID (Experimental): Participants received FSC 100/50 microgram (mcg) one inhalation as a combination product via DISKUS, twice daily in morning after awakening and in evening for up to 28 days
  Interventions: Drug: Fluticasone propionate/salmeterol
- FP 100 mcg BID (Experimental): Participants received FP 100 mcg one inhalation via DISKUS, twice daily in morning after awakening and in evening for up to 28 days.
  Interventions: Drug: Fluticasone Propionate

INTERVENTIONS:
Drug: Fluticasone propionate/salmeterol — Fluticasone propionate/salmeterol
  Arms: FSC 100/50 mcg BID
Drug: Fluticasone Propionate — Fluticasone Propionate
  Arms: FP 100 mcg BID

SUMMARY:
During this study, your child will need to attend up to 5 office visits and maintain regular telephone contact with the clinic. Certain office visits will include physical exams, medical history review, exercise challenge test (walking/running on a treadmill), electrocardiogram (ECG) tests, and lung function tests. All study related medications and medical examinations are provided at no cost. All study drugs are currently available by prescription to patients 4 years and older.

ELIGIBILITY:
Inclusion criteria:

* Diagnosed with persistent asthma for 3 months or longer.
* Experienced worsened asthma symptoms during physical activity.
* Using an inhaled steroid for the previous 4 weeks or longer (such as Aerobid, Azmacort, Flovent, Pulmicort, QVAR, and Vanceril).

Exclusion criteria:

* Used systemic steroids as either liquids, pills, or injections to treat asthma within the previous 3 months.
* Have only intermittent, seasonal, or exercise-induced asthma, and not persistent asthma.
* Admitted to a hospital within the previous 6 months due to asthma symptoms.
* Any poorly controlled medical conditions that may make study participation unsafe or inappropriate in the opinion of the study physician (such as cystic fibrosis, congenital heart disease, insulin dependent diabetes, glaucoma, drug allergies, etc.)
* The study physician will evaluate other medical criteria.

Ages: 4 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 248 (Actual)
Dates: Start 2003-12-23 (Actual); Primary Completion 2006-04-01 (Actual); Study Completion 2006-04-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (48):
- United States (48):
  - GSK Investigational Site, Little Rock, Arkansas
  - GSK Investigational Site, Huntington Beach, California
  - GSK Investigational Site, Orange, California
  - GSK Investigational Site, Palmdale, California
  - GSK Investigational Site, Paramount, California
  - GSK Investigational Site, San Diego, California
  - GSK Investigational Site, Torrance, California
  - GSK Investigational Site, Walnut Creek, California
  - GSK Investigational Site, Centennial, Colorado
  - GSK Investigational Site, Englewood, Colorado
  - GSK Investigational Site, Lakewood, Colorado
  - GSK Investigational Site, Miami, Florida
  - GSK Investigational Site, Tallahassee, Florida
  - GSK Investigational Site, Lilburn, Georgia
  - GSK Investigational Site, Chicago, Illinois
  - GSK Investigational Site, Hoffman Estates, Illinois
  - GSK Investigational Site, Metairie, Louisiana
  - GSK Investigational Site, Baltimore, Maryland
  - GSK Investigational Site, Glen Burnie, Maryland
  - GSK Investigational Site, North Dartmouth, Massachusetts
  - GSK Investigational Site, Minneapolis, Minnesota
  - GSK Investigational Site, Papillion, Nebraska
  - GSK Investigational Site, Skillman, New Jersey
  - GSK Investigational Site, Summit, New Jersey
  - GSK Investigational Site, Commack, New York
  - GSK Investigational Site, Utica, New York
  - GSK Investigational Site, Canton, Ohio
  - GSK Investigational Site, Cincinnati, Ohio
  - GSK Investigational Site, Dayton, Ohio
  - GSK Investigational Site, Gresham, Oregon
  - GSK Investigational Site, Medford, Oregon
  - GSK Investigational Site, Portland, Oregon
  - GSK Investigational Site, Erie, Pennsylvania
  - GSK Investigational Site, Hershey, Pennsylvania
  - GSK Investigational Site, Philadelphia, Pennsylvania
  - GSK Investigational Site, Pittsburgh, Pennsylvania
  - GSK Investigational Site, Charleston, South Carolina
  - GSK Investigational Site, Mt. Pleasant, South Carolina
  - GSK Investigational Site, Orangeburg, South Carolina
  - GSK Investigational Site, Dyersburg, Tennessee
  - GSK Investigational Site, Knoxville, Tennessee
  - GSK Investigational Site, Dallas, Texas
  - GSK Investigational Site, Houston, Texas
  - GSK Investigational Site, Murray, Utah
  - GSK Investigational Site, Richmond, Virginia
  - GSK Investigational Site, Greenfield, Wisconsin
  - GSK Investigational Site, Madison, Wisconsin
  - GSK Investigational Site, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] Pearlman D, Qaqundah P, Matz J, Yancey SW, Stempel DA, Ortega HG. Fluticasone propionate/salmeterol and exercise-induced asthma in children with persistent asthma. Pediatr Pulmonol. 2009 May;44(5):429-35. doi: 10.1002/ppul.20962. PMID 19382218
- See also: http://www.findclinicalstudy.com — http://www.findclinicalstudy.com
- Available data/document: Individual Participant Data Set: SFA100314 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: SFA100314 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: SFA100314 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: SFA100314 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: SFA100314 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: SFA100314 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted from 23 December 2003 to 23 April 2006 across 51 sites in the United States (US) and a total of 248 participants were randomized.
Pre-assignment Details: Out of 789 participants screened, 389 participants were screen failures and 152 participants were Baseline failures.
Groups:
- FSC 100/50 mcg BID: Participants received Fluticasone Propionate/Salmeterol Combination (FSC) 100/50 micrograms (mcg) one inhalation as a combination product via DISKUS, twice daily in morning after awakening and in evening for up to 28 days
- FP 100 mcg BID: Participants received Fluticasone Propionate (FP) 100 mcg one inhalation via DISKUS, twice daily in morning after awakening and in evening for up to 28 days.
Period: Overall Study
Arm/Group | FSC 100/50 mcg BID | FP 100 mcg BID
Started | 124 | 124
Completed | 111 | 102
Not Completed | 13 | 22
Not completed — Adverse Event | 2 | 7
Not completed — Protocol Violation | 5 | 4
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Exacerbation | 2 | 2
Not completed — Discontinued by sponsor | 1 | 1
Not completed — Non-compliance | 1 | 3
Not completed — misrandomized | 1 | 1
Not completed — Expired drug use | 1 | 2
Not completed — Investigator discretion | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- FSC 100/50mcg BID: Participants received FSC 100/50 mcg one inhalation as a combination product via DISKUS, twice daily in morning after awakening and in evening for up to 28 days.
- FP 100mcg BID: Participants received FP 100 mcg one inhalation via DISKUS, twice daily in morning after awakening and in evening for up to 28 days.
- Total: Total of all reporting groups
Arm/Group | FSC 100/50mcg BID | FP 100mcg BID | Total
Number analyzed (Participants) | 124 | 124 | 248
Age, Continuous [Mean (Standard Deviation); unit: Years] | 11.1 (3.33) | 11.0 (3.57) | 11.1 (3.45)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 49 | 50 | 99
  Male | 75 | 74 | 149
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Hispanic | 12 | 8 | 20
  Arabic/North African | 2 | 1 | 3
  Black | 26 | 29 | 55
  East & South East Asian | 0 | 2 | 2
  Japanese | 1 | 0 | 1
  South Asian | 1 | 1 | 2
  White/Caucasian | 81 | 81 | 162
  Other | 1 | 2 | 3

OUTCOME MEASURES:

1. Primary Outcome: Maximal Percent Change in Forced Expiratory Volume in 1 Second (FEV1) Following Exercise Challenge at Week 4
Description: FEV1 is a measure of lung function and is defined as the maximal amount of air that can be forcefully exhaled in one second. Maximal percent change in FEV1 following exercise challenge was defined as the percent change from pre-exercise baseline FEV1 to the minimum FEV1 collected within one hour following exercise challenge. Maximal percent change in FEV1 following exercise challenge was mean maximal percent change from pre-exercise baseline compared between treatment groups at Treatment Week 4. FEV1 was measured 5, 10, 15, 30, and 60 minutes post-exercise. The minimum FEV1 measured across these time points, regardless of any missing time points, will be used for the calculation of maximal percent change.
Time Frame: Baseline and Week 4
Population: Intent-to-Treat (ITT) population included all participants randomized to study drug. The number of participants available at that particular time point were used for analysis.
Measure: Mean (Standard Error); unit: Percent change
Arm/Group | FSC 100/50mcg BID | FP 100mcg BID
Number analyzed (Participants) | 113 | 104
Percent change | -9.5 (0.83) | -12.7 (1.06)
Statistical Analysis 1: Comparison: FSC 100/50mcg BID vs FP 100mcg BID; FSC 100/50mcg BID versus FP 100mcg BID for maximal percent change in FEV1 following exercise challenge at Week 4; Test type: Superiority or Other; p = 0.021, ANCOVA — LS Mean Difference, SE, CI, and p-value were from an ANCOVA model with terms for treatment, investigator, age stratum, and baseline value; Mean Difference (Net) = 3.0, 95% CI 2-sided [0.5 to 5.6], Standard Error of Mean 1.29 — LS Mean Diff was calculated as FSC 100/50mcg BID-FP 100mcg BID

2. Secondary Outcome: Four-hour Serial Post-dose FEV1 Area Under the Curve (AUC) on Treatment Day 1
Description: FEV1 AUC is mean AUC compared between treatment groups at Treatment Day 1. Baseline was defined as the pre-dose FEV1 measure from treatment Day 1. FEV1 AUC was calculated as the area of a trapezoid (calculated as the sum of the bases (top + bottom) divided by 2, then multiplied by width) above the baseline FEV1 area. For participants not completing a serial FEV1 measurement, the last observed post-dose FEV1 measurement was carried forward.
Time Frame: Immediately prior to dosing (0 time point), 30 minutes post-dose and 1, 2, 3, 4 hour post-dose on Day 1
Population: ITT population. Here, 'N' denotes participants with data available at the specified time point.
Measure: Mean (Standard Error); unit: Liters*hour
Arm/Group | FSC 100/50mcg BID | FP 100mcg BID
Number analyzed (Participants) | 119 | 120
Liters*hour | 0.70 (0.067) | 0.30 (0.059)
Statistical Analysis 1: Comparison: FSC 100/50mcg BID vs FP 100mcg BID; FSC 100/50mcg BID versus FP 100mcg BID for post-dose FEV1 AUC Day 1; Test type: Superiority or Other; p < 0.001, ANCOVA — LS Mean Diff, SE, CI, and p-value were from an ANCOVA model with terms for treatment, investigator, age stratum, and baseline value; Mean Difference (Net) = 0.41, 95% CI 2-sided [0.24 to 0.58], Standard Error of Mean 0.085 — LS Mean Diff was calculated as FSC 100/50mcg BID-FP 100mcg BID

3. Secondary Outcome: Change From Baseline in Morning Peak Expiratory Flow (AM PEF)
Description: PEF is defined as the maximum airflow during a forced expiration beginning with the lungs fully inflated. PEF was measured by the participants using a hand-held electronic peak flow meter each morning prior to the dose of study medication and any rescue albuterol/salbutamol inhalation aerosol use. Each participant was instructed to perform triplicate PEF measurements in the morning. Change from baseline was calculated as the endpoint value minus the baseline value. For AM PEF, baseline was defined as the average of the AM PEF values recorded on the day of Visit 2 (7-14 [+ or -4] days after Visit1) plus the 6 preceding days since AM PEF was measured in the morning.
Time Frame: Baseline and Up to Week 4
Population: ITT population. Here, 'N' denotes participants with data available at the specified time point.
Measure: Mean (Standard Error); unit: Liters/minute (L/min)
Arm/Group | FSC 100/50mcg BID | FP 100mcg BID
Number analyzed (Participants) | 117 | 113
Liters/minute (L/min) | 16.3 (2.99) | 9.1 (3.86)
Statistical Analysis 1: Comparison: FSC 100/50mcg BID vs FP 100mcg BID; FSC 100/50mcg BID versus FP 100mcg BID for AM PEF; Test type: Superiority or Other; p = 0.097, ANCOVA — LS Mean Diff, SE, CI, and p-values were from an ANCOVA model with terms for treatment, investigator, age stratum, and baseline value; Mean Difference (Net) = 8.1, 95% CI 2-sided [-1.5 to 17.6], Standard Error of Mean 4.83 — LS Mean Diffs were calculated as FSC 100/50mcg BID-FP 100mcg BID

4. Secondary Outcome: Change From Baseline in Evening (PM) PEF
Description: PEF is defined as the maximum airflow during a forced expiration beginning with the lungs fully inflated. PEF was measured by the participants using a hand-held electronic peak flow meter each evening prior to the dose of study medication after the symptom measurement and any rescue albuterol/salbutamol inhalation aerosol use. Each participant was instructed to perform triplicate PEF measurements in the evening. Change from baseline was calculated as the endpoint value minus the baseline value. Baseline was defined as the average of the values from the 7 days preceding Visit 2 (7-14 [+ or -4] days after Visit1) since these measures were derived from data collected in the evening.
Time Frame: Baseline and up to Week 4
Population: ITT population. Here, 'N' denotes participants with data available at the specified time point.
Measure: Mean (Standard Error); unit: L/min
Arm/Group | FSC 100/50mcg BID | FP 100mcg BID
Number analyzed (Participants) | 118 | 114
L/min | 10.8 (2.96) | 7.6 (3.03)
Statistical Analysis 1: Comparison: FSC 100/50mcg BID vs FP 100mcg BID; FSC 100/50mcg BID versus FP 100mcg BID PM PEF; Test type: Superiority or Other; p = 0.396, ANCOVA — [p-value comment as in outcome 3, analysis 1]; Mean Difference (Net) = 3.7, 95% CI 2-sided [-4.8 to 12.1], Standard Error of Mean 4.30 — LS Mean Diffs were calculated as FSC 100/50mcg BID-FP 100mcg BID

5. Secondary Outcome: Percent of Rescue-free Days
Description: A rescue-free day was defined as a day when no supplemental albuterol was taken (i.e., 0 puffs recorded for both AM and PM assessments of albuterol use in the daily diary). Percent of rescue-free days was calculated as the number of rescue-free days, divided by the total number of days in the treatment period, multiplied by 100 for each participant.
Time Frame: Up to Week 4
Population: ITT population. Here, 'N' denotes participants with data available at the specified time point.
Measure: Mean (Standard Error); unit: Percentage of days
Arm/Group | FSC 100/50mcg BID | FP 100mcg BID
Number analyzed (Participants) | 122 | 121
Percentage of days | 59.4 (3.21) | 54.7 (3.40)

6. Secondary Outcome: Percent of Symptom-free Days
Description: A symptom-free day was defined as a day with no symptoms (i.e., a score of 0, indicating no asthma symptoms during the day or previous night, recorded in the daily diary). Percent of symptom-free days was calculated as the number of symptom-free days, divided by the total number of days in the treatment period, multiplied by 100 for each participant.
Time Frame: Up to Week 4
Population: ITT population. Here, 'N' denotes participants with data available at the specified time point.
Measure: Mean (Standard Error); unit: Percentage of days
Arm/Group | FSC 100/50mcg BID | FP 100mcg BID
Number analyzed (Participants) | 122 | 121
Percentage of days | 27.3 (3.10) | 28.6 (3.04)

7. Secondary Outcome: Change From Baseline in Pediatric Asthma Quality of Life Questionnaire (PAQLQ)
Description: PAQLQ measures functional problems that are most troublesome to children with asthma. PAQLQ has 23 questions in 3 domains (activity limitation=5, emotional function=8, symptoms=10). Participants responded to each question on a 7-point scale (7= not bothered at all and 1= extremely bothered). The overall PAQLQ score is the mean of all 23 responses (minimum score 1= 5+8+10/23 and maximum score 7= 35+56+70/23) and the individual domain scores are the means of the items in those domains (minimum: 5/5, 8/8, 10/10 and maximum: 35/5, 56/8, 70/10). Minimum possible value is 1 (maximum impairment); maximum possible value is 7 (no impairment). Endpoint was defined from the last questionnaire collected during the double-blind treatment period or discontinuation visit (up to Week 4).
Time Frame: Baseline (Week 0) and up to Week 4
Population: ITT Population. The PAQLQ was administered only to participants >=7 years old.
Measure: Mean (Standard Error); unit: Scores on a scale
Arm/Group | FSC 100/50mcg BID | FP 100mcg BID
Number analyzed (Participants) | 104 | 102
Scores on a scale
  Activity limitation week 2: number analyzed (Participants) | 98 | 94
  Activity limitation week 2 | 0.78 (0.092) | 0.63 (0.100)
  Activity limitation week 4: number analyzed (Participants) | 89 | 79
  Activity limitation week 4 | 0.93 (0.113) | 0.75 (0.116)
  Activity limitation endpoint: number analyzed (Participants) | 103 | 101
  Activity limitation endpoint | 0.89 (0.104) | 0.67 (0.105)
  Emotional function Week 2: number analyzed (Participants) | 98 | 94
  Emotional function Week 2 | 0.44 (0.066) | 0.48 (0.089)
  Emotional function Week 4: number analyzed (Participants) | 89 | 79
  Emotional function Week 4 | 0.56 (0.096) | 0.47 (0.097)
  Emotional function endpoint: number analyzed (Participants) | 103 | 101
  Emotional function endpoint | 0.53 (0.090) | 0.42 (0.088)
  Symptoms Week 2: number analyzed (Participants) | 98 | 94
  Symptoms Week 2 | 0.39 (0.085) | 0.49 (0.081)
  Symptoms Week 4: number analyzed (Participants) | 89 | 79
  Symptoms Week 4 | 0.52 (0.101) | 0.55 (0.109)
  Symptoms Endpoint: number analyzed (Participants) | 103 | 101
  Symptoms Endpoint | 0.48 (0.094) | 0.51 (0.101)
  Overall score Week 2: number analyzed (Participants) | 98 | 94
  Overall score Week 2 | 0.49 (0.068) | 0.52 (0.074)
  Overall score Week 4: number analyzed (Participants) | 89 | 79
  Overall score Week 4 | 0.62 (0.091) | 0.57 (0.092)
  Overall score Endpoint: number analyzed (Participants) | 103 | 101
  Overall score Endpoint | 0.59 (0.084) | 0.51 (0.084)
Statistical Analysis 1: Comparison: FSC 100/50mcg BID vs FP 100mcg BID; FSC 100/50mcg BID versus FP 100mcg BID for activity limitation at Week 2; Test type: Superiority or Other; p = 0.168, ANCOVA — [p-value comment as in outcome 3, analysis 1]; Mean Difference (Net) = 0.18, 95% CI 2-sided [-0.08 to 0.43], Standard Error of Mean 0.129
Statistical Analysis 2: Comparison: FSC 100/50mcg BID vs FP 100mcg BID; FSC 100/50mcg BID versus FP 100mcg BID for activity limitation at Week 4; Test type: Superiority or Other; p = 0.465, ANCOVA — [p-value comment as in outcome 3, analysis 1]; Mean Difference (Net) = 0.11, 95% CI 2-sided [-0.18 to 0.40], Standard Error of Mean 0.147
Statistical Analysis 3: Comparison: FSC 100/50mcg BID vs FP 100mcg BID; FSC 100/50mcg BID versus FP 100mcg BID for activity limitation at Endpoint; Test type: Superiority or Other; p = 0.222, ANCOVA — LS Mean Diff, SE, CI, and p-values are from an ANCOVA model with terms for treatment, investigator, age stratum, and baseline value; Mean Difference (Net) = 0.16, 95% CI 2-sided [-0.10 to 0.42], Standard Error of Mean 0.133
Statistical Analysis 4: Comparison: FSC 100/50mcg BID vs FP 100mcg BID; FSC 100/50mcg BID versus FP 100mcg BID for emotional function at Week 2; Test type: Superiority or Other; p = 0.294, ANCOVA — [p-value comment as in outcome 3, analysis 1]; Mean Difference (Net) = -0.10, 95% CI 2-sided [-0.29 to 0.09], Standard Error of Mean 0.096
Statistical Analysis 5: Comparison: FSC 100/50mcg BID vs FP 100mcg BID; FSC 100/50mcg BID versus FP 100mcg BID for emotional function at Week 4; Test type: Superiority or Other; p = 0.828, ANCOVA — [p-value comment as in outcome 3, analysis 1]; Mean Difference (Net) = -0.02, 95% CI 2-sided [-0.24 to 0.19], Standard Error of Mean 0.111
Statistical Analysis 6: Comparison: FSC 100/50mcg BID vs FP 100mcg BID; FSC 100/50mcg BID versus FP 100mcg BID for emotional function at Endpoint; Test type: Superiority or Other; p = 0.903, ANCOVA — [p-value comment as in outcome 3, analysis 1]; Mean Difference (Net) = 0.01, 95% CI 2-sided [-0.19 to 0.22], Standard Error of Mean 0.103
Statistical Analysis 7: Comparison: FSC 100/50mcg BID vs FP 100mcg BID; FSC 100/50mcg BID versus FP 100mcg BID for symptoms at Week 2; Test type: Superiority or Other; p = 0.464, ANCOVA; LS Mean Diff, SE, CI, and p-values were from an ANCOVA model with terms for treatment, investigator, age stratum, and baseline value; Mean Difference (Net) = -0.08, 95% CI 2-sided [-0.30 to 0.14], Standard Error of Mean 0.112
Statistical Analysis 8: Comparison: FSC 100/50mcg BID vs FP 100mcg BID; FSC 100/50mcg BID versus FP 100mcg BID for symptoms at Week 4; Test type: Superiority or Other; p = 0.551, ANCOVA — [p-value comment as in outcome 3, analysis 1]; Mean Difference (Net) = -0.07, 95% CI 2-sided [-0.32 to 0.17], Standard Error of Mean 0.124
Statistical Analysis 9: Comparison: FSC 100/50mcg BID vs FP 100mcg BID; FSC 100/50mcg BID versus FP 100mcg BID for symptoms at Endpoint; Test type: Superiority or Other; p = 0.633, ANCOVA — [p-value comment as in outcome 3, analysis 1]; Mean Difference (Net) = -0.06, 95% CI 2-sided [-0.30 to 0.18], Standard Error of Mean 0.123
Statistical Analysis 10: Comparison: FSC 100/50mcg BID vs FP 100mcg BID; FSC 100/50mcg BID versus FP 100mcg BID for overall score at Week 2; Test type: Superiority or Other; p = 0.700, ANCOVA — [p-value comment as in outcome 7, analysis 3]; Mean Difference (Net) = -0.04, 95% CI 2-sided [-0.22 to 0.15], Standard Error of Mean 0.094
Statistical Analysis 11: Comparison: FSC 100/50mcg BID vs FP 100mcg BID; FSC 100/50mcg BID versus FP 100mcg BID for overall score at Week 4; Test type: Superiority or Other; p = 0.860, ANCOVA — [p-value comment as in outcome 3, analysis 1]; Mean Difference (Net) = -0.02, 95% CI 2-sided [-0.23 to 0.20], Standard Error of Mean 0.109
Statistical Analysis 12: Comparison: FSC 100/50mcg BID vs FP 100mcg BID; FSC 100/50mcg BID versus FP 100mcg BID for overall score at Endpoint; Test type: Superiority or Other; p = 0.919, ANCOVA — [p-value comment as in outcome 3, analysis 1]; Mean Difference (Net) = 0.01, 95% CI 2-sided [-0.19 to 0.21], Standard Error of Mean 0.103

ADVERSE EVENTS:
Time Frame: Adverse events and serious adverse events were collected from Visit 1 (Screening) until completion of the study (Up to 58 days)
Description: ITT population was used for the analysis of adverse events and serious adverse events.
Arm/Group | FSC 100/50mcg BID | FP 100mcg BID
All-Cause Mortality (participants affected / at risk) | 0/124 | 0/124
Serious Adverse Events (participants affected / at risk) | 0/124 | 0/124
Other Adverse Events (participants affected / at risk) | 37/124 | 35/124
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | FSC 100/50mcg BID (N=124) | FP 100mcg BID (N=124)
Upper respiratory tract infection (Infections and infestations) | 4 | 2
Nasopharyngitis (Infections and infestations) | 2 | 1
Bronchitis (Infections and infestations) | 0 | 2
Gastroenteritis (Infections and infestations) | 2 | 0
Gastroenteritis viral (Infections and infestations) | 1 | 1
Pharyngitis (Infections and infestations) | 1 | 1
Pharyngitis streptococcal (Infections and infestations) | 1 | 1
Viral upper respiratory tract infection (Infections and infestations) | 0 | 2
Fungal infection (Infections and infestations) | 0 | 1
Herpes simplex (Infections and infestations) | 1 | 0
Oral candidiasis (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 0 | 1
Sinusitis (Infections and infestations) | 0 | 1
Tinea pedis (Infections and infestations) | 0 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Abdominal pain upper (Gastrointestinal disorders) | 3 | 2
Nausea (Gastrointestinal disorders) | 2 | 1
Anal fissure (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 0
Tooth impacted (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0
Headache (Nervous system disorders) | 4 | 6
Dizziness (Nervous system disorders) | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 4
Rash (Skin and subcutaneous tissue disorders) | 1 | 2
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 | 0
Eczema (Skin and subcutaneous tissue disorders) | 0 | 1
Pityriasis rosea (Skin and subcutaneous tissue disorders) | 1 | 0
Skin laceration (Injury, poisoning and procedural complications) | 1 | 1
Contusion (Injury, poisoning and procedural complications) | 0 | 1
Excoriation (Injury, poisoning and procedural complications) | 0 | 1
Eye injury (Injury, poisoning and procedural complications) | 0 | 1
Foot fracture (Injury, poisoning and procedural complications) | 0 | 1
Joint sprain (Injury, poisoning and procedural complications) | 1 | 0
Pyrexia (General disorders) | 2 | 1
Chest pain (General disorders) | 1 | 0
Irritability (General disorders) | 1 | 0
Cerumen impaction (Ear and labyrinth disorders) | 0 | 1
Middle ear effusion (Ear and labyrinth disorders) | 0 | 1
Food allergy (Immune system disorders) | 1 | 0
Increased appetite (Metabolism and nutrition disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Asperger's disorder (Psychiatric disorders) | 0 | 1
Tongue tie operation (Surgical and medical procedures) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.